CLINICAL TRIAL: NCT07292259
Title: The Efficacy of Combined Thalidomide and Hydroxyurea Therapy in Transfusion Dependent β-thalassemia (TDBT), Phase II Trial
Brief Title: Combination of Thalidomide and Hydroxyuria in Transfusion Dependent Thalasemmia
Acronym: Thal-H
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pakistan Blood and Marrow Transplant (PBMT) Group (Other)
Responsible Party: Principal Investigator, Professor Tariq Ghafoor, Director AFBMTC, Pakistan Blood and Marrow Transplant (PBMT) Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBMT-1; 6871 (Other: AFBMTC)
Record Dates: First submitted 2025-11-13; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Transfusion Dependent Beta Thalassemia
Keywords: Thalidomide, Hydoxyurea, Transfusion dependent thalassemia
MeSH Terms: interventions — Hydroxyurea; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A combination of thalidomide and hydroxyurea is added to patients diagnosed with TDT (Experimental): * The trial include Hydroxyurea (HU) and Thalidomide in combination. The starting dose of Hydroxyurea will be 20 mg/kg once daily and of thalidomide will be 2.5-3 mg/kg once a day adjusted to nearest multiple of 10, at bedtime. Among those with partial response (PR) or no response (NR) after two months, the dose of thalidomide will be escalated in increments of 1 mg/kg/day at four weeks interval to a maximum of 5 mg/kg/day (maximum dose 100 mg/day).
  * To prevent thrombosis, aspirin (2-4 mg/kg per day) will be used. All patients will receive Folic acid 2 to 5 mg once daily.
  Interventions: Drug: ADDITION OF THALIDOMIDE AND HYDROXYUREA

INTERVENTIONS:
Drug: ADDITION OF THALIDOMIDE AND HYDROXYUREA — The intervention includes Hydroxyurea (HU) and Thalidomide in combination. The starting dose of Hydroxyurea will be 20 mg/kg once daily and of thalidomide will be 2.5-3 mg/kg once a day adjusted to nearest multiple of 10, at bedtime. Among those with partial response (PR) or no response (NR) after two months, the dose of thalidomide will be escalated in increments of 1 mg/kg/day at four weeks interval to a maximum of 5 mg/kg/day (maximum dose 100 mg/day).
  * To prevent thrombosis, aspirin (2-4 mg/kg per day) will be used. All patients will receive Folic acid 2 to 5 mg once daily.
  * Patients will also continue the iron chelation therapy (Deferasirox, Deferiprone or Deferoxamine) in case of iron overload.
  Other Names: Hydrea and Thalidomide

SUMMARY:
Beta thalassemia Major (BTM) is the most common hemoglobinopathy caused by mutations in the beta-globin gene . Worldwide, approximately 80 million people carry thalassemia gene mutation. Around 23,000 babies are affected by BTM each year, of which around 90% belong to low- or middle-income nations.

In Pakistan, the carrier prevalence of thalassemia is 5-7% resulting in a significant population of approximately 10 million carriers in the general population. There are 50,000 thalassemia patients registered in treatment facilities around the country, one of the highest global prevalence rates for transfusion dependent BTM. The average life expectancy of BTM patients in Pakistan is around 10 years of age, while life expectancy in developed countries is around 50 to 60 years. This difference is due to poor transfusion support, transfusion-transmitted infections (TTIs) and inadequate iron chelation leading to hepatotoxicity and cardiac failure.

The standard of care for BTM remains bone marrow transplantation or lifelong blood transfusions followed by iron chelation therapies. While standard care involves, challenges such as limited resources, lack of access to transplant services, and transfusion-related complications persist, particularly in low-and-middle-income countries.

DETAILED DESCRIPTION:
Beta thalassemia Major (BTM) is the most common hemoglobinopathy caused by mutations in the beta-globin gene . Worldwide, approximately 80 million people carry thalassemia gene mutation. Around 23,000 babies are affected by BTM each year, of which around 90% belong to low- or middle-income nations.

In Pakistan, the carrier prevalence of thalassemia is 5-7% resulting in a significant population of approximately 10 million carriers in the general population. There are 50,000 thalassemia patients registered in treatment facilities around the country, one of the highest global prevalence rates for transfusion dependent BTM. The average life expectancy of BTM patients in Pakistan is around 10 years of age, while life expectancy in developed countries is around 50 to 60 years. This difference is due to poor transfusion support, transfusion-transmitted infections (TTIs) and inadequate iron chelation leading to hepatotoxicity and cardiac failure.

The standard of care for BTM remains bone marrow transplantation or lifelong blood transfusions followed by iron chelation therapies. While standard care involves, challenges such as limited resources, lack of access to transplant services, and transfusion-related complications persist, particularly in low-and-middle-income countries.

Hydroxyurea (HU), an FDA-approved inducer of fetal hemoglobin (HbF), has shown promise in reducing or eliminating the need for frequent blood transfusions in β-thalassemia patients. However, a subset of patients exhibits limited responsiveness to HU, necessitating exploration of adjunct or alternative therapies. Thalidomide, an immune modulator, has demonstrated transfusion reduction by suppressing nuclear factor-κB induction, potentially increasing HbF levels.

The primary aim of this prospective study is to determine the efficacy of the combination of thalidomide and hydroxyurea in reducing transfusion frequency in patients with β-thalassemia Major. The secondary objectives are to document the spectrum of significant adverse drug reactions as well to document any alteration in the spleen size and serum ferritin levels.

ELIGIBILITY:
Inclusion Criteria:

• Patients suffering from Transfusion Dependent β-thalassemia (TDBT) more than two years of age of either sex will be included in the study.

Exclusion Criteria:

* Age less than two years.
* Patients having cardiac, hepatic, pulmonary, renal or neurological dysfunction or history of thrombosis.
* Both male and female participants of childbearing potential will be excluded due to the teratogenicity of thalidomide.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Red Blood Cell Transfusions after starting a combination of Thalidomide and hydroxyurea | 01 Year
  The frequency of Red Blood cell transfusions before the start of intervention will be noted. At 03 months, 06 months, and 12 months of intervention (Thalidomide and hydroxyurea) number of Red Blood cell transfusions will be documented.

SECONDARY OUTCOMES:
To document the spectrum and frequency of significant adverse drug reactions. | 01 Year
  Monitoring and recording any adverse effects associated with thalidomide and hydroxyurea therapy at Day-90, Day-180, and Day-365.
  Patients will be contacted on the telephone weekly by the drug safety monitoring board and will be screened for any side effects of the intervention.
To assess changes in spleen size during the intervention. | 01 Year
  Assessment of spleen size in centimeters at Day-01, Day-90, Day-180, and Day-365 of intervention.
Monitoring of Serum Ferritin levels in ng/ml during the time of intervention. | 01 Year
  Measurement of Serum Ferritin Levels in ng/ml at Day-01, Day-90, Day-180, and Day-365.

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Ghafoor, FCPS,FRCP, Study Director — National Institute of Blood and Marrow Transplant (NIBMT), Pakistan
Locations (7):
- Pakistan (7):
  - Armed Forces Bone Marrow Transplant Center, Islamabad, Punjab Province
  - Armed Forces Bone Marrow Transplant Center, Rawalpindi, Punjab Province
  - AFBMTC (Clinical Trial and Research Cell), Rawalpindi, Punjab Province
  - AFBMTC (CT&RC), CMH Medical Complex, Rawalpindi, Punjab Province
  - AFBMTC (CT&RC), Medical Complex, Rawalpindi, Punjab Province
  - AFBMTC, CMH Medical Complex, Rawalpindi, Punjab Province
  - Armed Forces Bone Marrow Transplant Center Rawalpindi Pakistan, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: Yes
The investigators may share de-identified IPD upon reasonable request, beginning 9 months after publication and available for up to 24 months, following review and data-sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Six months after completion of study
Access Criteria: Contact with PI
URL: https://pbmt.org.pk/

REFERENCES:
- [Result] Li X, Hu S, Liu Y, Huang J, Hong W, Xu L, Xu H, Fang J. Efficacy of Thalidomide Treatment in Children With Transfusion Dependent beta-Thalassemia: A Retrospective Clinical Study. Front Pharmacol. 2021 Aug 12;12:722502. doi: 10.3389/fphar.2021.722502. eCollection 2021. PMID 34456732
- [Result] Garg A, Patel K, Shah K, Trivedi D, Raj A, Yadav R, Shah S. Safety and Efficacy of Thalidomide and Hydroxyurea Combination in Beta Thalassemia Patients. Indian J Hematol Blood Transfus. 2023 Jan;39(1):85-89. doi: 10.1007/s12288-022-01536-y. Epub 2022 Apr 21. PMID 36699430
- [Result] Chen J, Zhu W, Cai N, Bu S, Li J, Huang L. Thalidomide induces haematologic responses in patients with beta-thalassaemia. Eur J Haematol. 2017 Nov;99(5):437-441. doi: 10.1111/ejh.12955. Epub 2017 Sep 27. PMID 28850716
- [Result] Nag A, Radhakrishnan VS, Kumar J, Bhave S, Mishra DK, Nair R, Chandy M. Thalidomide in Patients with Transfusion-Dependent E-Beta Thalassemia Refractory to Hydroxyurea: A Single-Center Experience. Indian J Hematol Blood Transfus. 2020 Apr;36(2):399-402. doi: 10.1007/s12288-020-01263-2. Epub 2020 Mar 2. PMID 32425398
- [Result] Ansari SH, Ansari I, Wasim M, Sattar A, Khawaja S, Zohaib M, Hussain Z, Adil SO, Ansari AH, Ansari UH, Farooq F, Masqati NU. Evaluation of the combination therapy of hydroxyurea and thalidomide in beta-thalassemia. Blood Adv. 2022 Dec 27;6(24):6162-6168. doi: 10.1182/bloodadvances.2022007031. PMID 35477175